CLINICAL TRIAL: NCT03120949
Title: A Multicenter, Open-Label, Phase III Study of the Efficacy and Safety of Olokizumab in Subjects With Moderately to Severely Active Rheumatoid Arthritis
Brief Title: Efficacy and Safety of Olokizumab in Subjects With Moderately to Severely Active Rheumatoid Arthritis
Acronym: CREDO 4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: R-Pharm International, LLC (Industry)
Collaborators: IQVIA Pvt. Ltd (Industry); OCT Clinical Trials (Other)
Responsible Party: Sponsor
Organization: R-Pharm (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL04041024; 2015-005309-35 (EudraCT Number)
Record Dates: First submitted 2017-02-07; First posted 2017-04-19 (Actual); Results first posted 2022-06-07 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; moderate; severe; subcutaneous; Olokizumab; open-label
MeSH Terms: conditions — Arthritis, Rheumatoid; Lymphoma, Follicular | interventions — olokizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm 1: OKZ 64 mg q4w + MTX (Experimental): Olokizumab 64 mg SC q4w + concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular).
  Interventions: Drug: Olokizumab 64 mg SC q4w; Drug: Concomitant treatment
- Treatment Arm 2: OKZ 64 mg q2w + MTX (Experimental): Olokizumab 64 mg SC q2w + concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular).
  Interventions: Drug: Olokizumab 64 mg SC q2w; Drug: Concomitant treatment

INTERVENTIONS:
Drug: Olokizumab 64 mg SC q4w — 160 mg/mL sterile solution for SC injection in a 2 mL clear Type I glass vial with target volume of 0.4 mL or in the pre-filled syringe (PFS).PFS is composed of a 1 mL clear Type I glass barrel vial with target volume of 0.4 mL.
  Arms: Treatment Arm 1: OKZ 64 mg q4w + MTX
Drug: Olokizumab 64 mg SC q2w — 160 mg/mL sterile solution for SC injection in a 2 mL clear Type I glass vial with target volume of 0.4 mL or in the pre-filled syringe (PFS). PFS is composed of a 1 mL clear Type I glass barrel vial with target volume of 0.4 mL.
  Arms: Treatment Arm 2: OKZ 64 mg q2w + MTX
Drug: Concomitant treatment — Methotrexate 15 to 25 mg/week (or ≥ 10 mg/week if there was documented intolerance to higher doses). (Subject maintained their stable dose and route (oral, SC, or IM) during the core study and for ≥ 12 additional weeks of OLE.)
  Folic acid ≥ 5 mg per week or equivalent

SUMMARY:
The primary objective of this study was to evaluate the long-term safety and tolerability of olokizumab (OKZ) 64 mg administered subcutaneously (SC) once every 2 weeks (q2w) or once every 4 weeks (q4w) in subjects with moderately to severely active rheumatoid arthritis (RA) who previously had completed 24 weeks of double-blind treatment in Study CREDO 1, 2 or 3 (core studies). The long-term efficacy, immunogenicity, the physical function and quality of life of subjects received long-term treatment with OKZ were assessed as well.

DETAILED DESCRIPTION:
This OLE study (CL04041024) included an 82-week open-label Treatment Period that followed completion of one of the core studies (Study CREDO 1, 2 or 3). The OLE open-label Treatment Period lasted from Visit 1 (OLE Baseline/Week 24) to Visit 10 (End of Treatment (EoT)/Week 106), followed by a 20-week Safety Follow-Up Period from Week 106 to Week 126. The first visit of the OLE study was the same visit as the Week 24 visit in the core studies.

Subjects were randomized to 1 of the 2 OKZ treatment groups in the OLE study based on the treatment received in the core studies. Subjects who had received OKZ (q2w or q4w) in the core study in which they had participated (including subjects who received placebo in Study CREDO 3 and were re-randomized to OKZ at Week 16) received the same OKZ treatment regimen in the OLE study. Subjects who had received placebo (Study CREDO 1 and CREDO 2) or adalimumab (Study CREDO 2) in the core study in which they had participated were randomized in a 1:1 ratio to OKZ 64 mg q2w or OKZ 64 mg q4w regimens in the OLE study.

For the first 12 weeks of the OLE, all subjects were required to remain on a stable dose of background methotrexate (MTX) at 15 to 25 mg/week (or≥10 mg/week if there was documented intolerance to higher doses) with a stable route of administration (oral, SC, or intramuscular (IM)). After 12 weeks (Visit 4 [Week 36] of the OLE study), the Investigator might adjust the MTX dosage and route, per local guidelines. Methotrexate might be adjusted only for safety reasons according to Investigator discretion before Visit 4 (Week 36) of the OLE study.

Subjects who had been on rescue disease-modifying anti-rheumatic drugs (DMARDs) during the core studies were asked to continue these medications for the first 12 weeks of the OLE study. The Investigator could adjust these background medications if deemed appropriate after Visit 4 (Week 36) of the OLE study. Background rescue therapy might be adjusted only for safety reasons according to Investigator discretion before Visit 4 (Week 36) of the OLE study.

Throughout the study, concomitant treatment with folic acid ≥ 5 mg per week or equivalent was required for all subjects.

Subjects returned to the study site periodically for safety and response assessments as per the Schedule of Events.

The last dose of open-label study treatment in the OLE study was administered at Week 104 for all subjects. After completion of the 82-week open-label Treatment Period, subjects entered the 20-week Safety Follow-Up Period. During the Safety Follow-Up Period, subjects returned for 3 visits at +4, +8, and +22 weeks after the last dose of study treatment.

Subjects who discontinued the open-label treatment prematurely required to come for the EoT Visit 2 weeks after the last study treatment administration and then return for the 3 Safety Follow-Up Visits +4, +8, and +22 weeks after the last study treatment administration.

Adverse events were assessed throughout the study period and evaluated using the Common Technology Criteria version 4.0 (CTCAE v 4.0).

There were ongoing monitoring of safety events, including laboratory findings by the Sponsor or its designee. In addition, safety parameters were assessed throughout the study by an independent Data Safety Monitoring Board (DSMB).

ELIGIBILITY:
Inclusion Criteria:

Subjects may be enrolled in the study only if they meet all of the following criteria:

1. Subject must be willing and able to sign informed consent
2. Subject must have completed the 24-week double-blind Treatment Period in 1 of the 3 core studies (CL04041022, CL04041023, or CL04041025).
3. Subject must have maintained their stable dose (and route) of MTX 15 to 25 mg/week (or ≥ 10 mg/week if there is documented intolerance to higher doses) during the core study and plan to maintain the same dose and route of administration for ≥ 12 additional weeks
4. Subjects must be willing to take folic acid or equivalent throughout the study.

Exclusion Criteria:

1. Subject with any medically important condition in the core study (e.g., clinically significant laboratory values, frequent Adverse events (AEs) or serious adverse events (SAEs), infection SAEs, and/or other concurrent severe and/or uncontrolled medical condition) which would make this subject unsuitable for inclusion in the open-label extension (OLE) study in the Investigator's judgement.
2. Subject has evidence of active tuberculosis (TB)
3. Subject with a positive or repeated indeterminate interferon-gamma release assay (IGRA) result at Week 22 of the core study

   - Subjects may be enrolled in the OLE study if they fulfill all 3 of the following criteria prior to the first dose of study treatment:
   1. Active TB is ruled out by a certified TB specialist or pulmonologist who is familiar with diagnosing and treating TB (as acceptable per local practice);
   2. The subject starts prophylaxis for latent TB infection (LTBI) according to country-specific/Centers for Disease Control and Prevention (CDC) guidelines (treatment with isoniazid for 6 months is not an appropriate prophylactic regime for this study and it should not be used); and
   3. The subject is willing to complete the entire course of recommended LTBI therapy.
4. Subject has planned surgery during the first 12 weeks of the OLE study
5. Female subjects who are pregnant or who are planning to become pregnant during the study or within 6 months of the last dose of study drug
6. Female subjects of childbearing potential (unless permanent cessation of menstrual periods, determined retrospectively after a woman has experienced 12 months of natural amenorrhea as defined by the amenorrhea with underlying status [e.g., correlative age] or 6 months of natural amenorrhea with documented serum follicle-stimulating hormone levels >40 mIU/mL and estradiol <20 pg/mL) who are not willing to use a highly effective method of contraception during the study and for at least 6 months after the last administration of study treatment OR Male subjects with partners of childbearing potential not willing to use a highly effective method of contraception during the study and for at least 3 months after the last administration of study treatment.

   Highly effective contraception is defined as:
   * Female sterilization surgery: hysterectomy, surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least 6 weeks prior to the first dose of study treatment in the core study

     * In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by documented follow-up hormone level assessment
   * Total abstinence if it is the preferred and constant lifestyle of the subject. Thus, periodic abstinence such as ovulation, symptothermal, postovulation, calendar methods, and withdrawal are not acceptable methods of contraception.
   * Male sterilization surgery: at least 6 months prior to the first dose of study treatment in the core study (with the appropriate postvasectomy documentation of the absence of sperm in the ejaculate). For female subjects, the vasectomized male should be the only partner.
   * Placement of established intrauterine device (IUD): IUD copper or IUD with progesterone
   * Barrier method (condom and intravaginal spermicide, cervical caps with spermicide, or diaphragm with spermicide) in combination with the following: established oral, injected, or implanted hormone methods of contraception or contraceptive patch.
7. Subject is unwilling or unable to follow the procedures outlined in the protocol.
8. Other medical or psychiatric conditions, or laboratory abnormalities that may increase the potential risk associated with study participation and administration of the study treatment, or that may affect study results interpretation and, as per Investigator's judgement, make the subject ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2106 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — Chief Medical Officer, R-Pharm
Locations (239):
- United States (71):
  - AZ Arthritis & Rheum' Research, Mesa, Arizona
  - Arizona Arthritis & Rheumatology Associates, P.C., Phoenix, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Sun City, Arizona
  - CHI St. Vincent Hot Springs, Hot Springs, Arkansas
  - Medvin Clinical Research, Covina, California
  - C.V Mehta MD Med Corp.., Hemet, California
  - Advanced Medical Research, LLC, La Palma, California
  - Valerius Medical Group, Los Alamitos, California
  - Stanford University School of Medicine, Palo Alto, California
  - Rheumatology Center of San Diego, San Diego, California
  - East Bay Rheumatology Medical Group, Inc., San Leandro, California
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - Center for Rheumatology Research, Comprehensive Rheumatology Center, West Hills, California
  - Medvin Clinical Research, Whittier, California
  - Denver Arthritis Clinic, Denver, Colorado
  - New England Research Associates LLC, Bridgeport, Connecticut
  - Javed Rheumatology Associates, Newark, Delaware
  - RASF - Clinical Research Center, Boca Raton, Florida
  - Reliable Clinical Research, LLC, Hialeah, Florida
  - Pharmax Research Clinic, Miami, Florida
  - Medical Research Center of Miami, Miami, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - Omega Research Consultants, Orlando, Florida
  - Arthritis Research of Florida, INC, Palm Harbor, Florida
  - Family Clinical Trials, LLC., Pembroke Pines, Florida
  - AdventHealth Medical Group, PA, Tampa, Florida
  - Lovelace Scientific Resources, Inc., Venice, Florida
  - Arthritis Center of North Georgia, Gainesville, Georgia
  - Marietta Rheumatology Associates, PC, Marietta, Georgia
  - Institute of Arthritis Research, Idaho Falls, Idaho
  - University of Kansas Hospital, Kansas City, Kansas
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - The Arthritis & Diabetes Clinic, Inc., Monroe, Louisiana
  - Klein and Associates, M.D., P.A., Hagerstown, Maryland
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - AA MRC LLC Ahmed Arif Medical Research Center, Grand Blanc, Michigan
  - North MS Medical Clinics, Inc., Tupelo, Mississippi
  - Glacier View Research Institute-Rheumatology, Kalispell, Montana
  - Physician Research Collaboration, Lincoln, Nebraska
  - Arthritis & Osteoporosis Associates, PA, Freehold, New Jersey
  - Lovelace Scientific Resources, Inc., Albuquerque, New Mexico
  - NYU Langone ambulatory care, Brooklyn, New York
  - Medication Management, LLC, Greensboro, North Carolina
  - Cape Fear Arthritis Care, Leland, North Carolina
  - Carolina Arthritis Associates, Wilmington, North Carolina
  - Trinity Medical Group, Minot, North Dakota
  - Cincinnati Rheumatic Disease Study Group, Cincinnati, Ohio
  - STAT Research, Inc., Dayton, Ohio
  - Clinical Research Source, Inc., Toledo, Ohio
  - Health Research of Oklahoma, PLLC, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, P.C., Duncansville, Pennsylvania
  - Arthritis Group, Philadelphia, Pennsylvania
  - Low Country Rheumatology, PA, Summerville, South Carolina
  - Amarillo Center for Clinical Research, Amarillo, Texas
  - Austin Regional Clinic, P.A., Austin, Texas
  - Accurate Clinical Management., LLC, Baytown, Texas
  - Precision Comprehensive Clinical Research Solutions, Colleyville, Texas
  - Pioneer Research Solutions, Inc., Cypress, Texas
  - Therapeutic Concepts Rheumatology,LLC, Houston, Texas
  - Rheumatology Clinic of Houston, P.A., Houston, Texas
  - Houston Institute For Clinical Research, Houston, Texas
  - Accurate Clinical Mangemnt - Partner, Houston, Texas
  - Accurate Clinical Research, Inc., Houston, Texas
  - Accurate Clinical Research, Inc., League City, Texas
  - West Texas Clinical Research, Lubbock, Texas
  - Dr Alex De Jesus Rheumatology, P.A., San Antonio, Texas
  - Advanced Rheumatology of Houston, The Woodlands, Texas
  - DM Clinical Research, Tomball, Texas
  - Arthritis Northwest, PLLC, Spokane, Washington
- Argentina (14):
  - Centro de Investigaciones Medicas Mar del Plata, Mar del Plata, Buenos Aires
  - Instituto Medico CER, Quilmes, Buenos Aires
  - Instituto de Investigaciones Clinicas Quilmes, Quilmes, Buenos Aires
  - Sanatorio San Martin, Venado Tuerto, Santa Fe Province
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán, Tucumán Province
  - Instituto de Investigaciones Clinicas-Mar del Plata, Buenos Aires
  - Organizacion Medica de Investigacion (OMI), Ciudad Autonoma Buenos Aires
  - APRILLUS Asistencia e Investigacion, Ciudad Autonoma Buenos Aires
  - Instituto Centenario, Ciudad Autonoma Buenos Aires
  - Hospital Privado Centro Medico de Cordoba, Córdoba
  - Instituto DAMIC Fundacion Rusculleda, Córdoba
  - CER San Juan Centro Polivalente de Asistencia e Inv. Clinica, San Juan
  - Centro de Investigaciones Reumatológicas, San Miguel de Tucumán
  - Clinica de Higado y Aparato Digestivo, Santa Fe
- Belarus (2):
  - Minsk City Clinical Hospital #1, Minsk, Minsk Oblast
  - Vitebsk Clinical Hospital, Vitebsk, Vitebsk Oblast
- Brazil (14):
  - HUWC - UFC - Hospital Universitário Walter Cantídio - Universidade Federal do Ceará, Fortaleza, Ceará
  - CEDOES - Diagnóstico e Pesquisa, Vitória, Espírito Santo
  - CIP - Centro Internacional de Pesquisa, Goiânia, Goiás
  - CMiP - Centro Mineiro de Pesquisa, Juiz de Fora, Minas Gerais
  - CETI - Centro de Estudos em Terapias Inovadoras Ltda., Curitiba, Paraná
  - Clinilive - Clínica do Idoso e Pesquisa Clínica, Maringá, Paraná
  - Hospital Bruno Born, Lajeado, Rio Grande do Sul
  - LMK Serviços Médicos S/S Ltda, Pôrto Alegre, Rio Grande do Sul
  - Clínica de Neoplasias Litoral Ltda., Itajaí, Santa Catarina
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Centro Multidisciplinar de Estudos Clínicos - CEMEC, São Bernardo do Campo, São Paulo
  - CCBR Brasil Centro de Pesquisas e Análises Clínicas Ltda., Rio de Janeiro
  - CPCLIN - Centro de Pesquisas Clínicas Ltda., São Paulo
  - Associação de Assistência à Criança Deficiente - AACD, São Paulo
- Bulgaria (12):
  - DCC 'Sv. Pantaleymon' OOD, Pleven
  - UMHAT Pulmed OOD, Plovdiv
  - UMHAT "Kaspela", EOOD, Plovdiv
  - MHAT - Ruse, AD, Rousse
  - Medizinski Zentar-1-Sevlievo EOOD, Sevlievo
  - MHAT - Shumen, AD, Shumen
  - NMTH "Tsar Boris III", Sofia
  - MHAT "Lyulin", EAD, Sofia
  - Medical Center "Excelsior", OOD, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia
  - MC "Synexus - Sofia", EOOD, Sofia
  - MDHAT 'Dr. Stefan Cherkezov', AD, Veliko Tarnovo
- Colombia (5):
  - Centro de Reumatologia y Ortopedia SAS, Barranquilla
  - Centro de Investigacion en Reumatologia y Especialidades Medicas SAS. CIREEM, Bogotá
  - Fundacion Instituto de Reumatologia Fernando Chalem, Bogotá
  - Medicity S.A.S., Bucaramanga
  - Clinica de Artritis Temprana S.A.S, Cali
- Czechia (19):
  - CCR Brno s.r.o, Brno
  - IMEDICA s.r.o., Brno
  - Revmatologie s.r.o., Brno
  - Nemocnice Jihlava p.o., Jihlava
  - MUDr Gabriela Simkova Ordinace Lekare Specialisty Interna Revmatologie, Kladno
  - CTCenter MaVe s.r.o., Olomouc
  - Vesalion s.r.o., Ostrava
  - ARTROSCAN s.r.o., Ostrava - Trebovice
  - ARTHROHELP s.r.o., Pardubice
  - CCR Czech, a.s., Pardubice
  - CLINTRIAL s.r.o., Prague
  - Revmatologicky ustav, Prague
  - CCR Prague s.r.o., Prague
  - MUDR Zuzana URBANOVA Revmatologie, Prague
  - Affidea Praha s.r.o., Prague
  - Fakultni nemocnice v Motole, Prague
  - MUDR Zuzana URBANOVA Revmatologie, Praha 4 Nusle
  - Medical Plus s.r.o., Uherské Hradiště
  - PV - MEDICAL, s.r.o., Zlín
- Estonia (2):
  - East Tallinn Central Hospital, Tallinn
  - Meditrials OU, Tartu
- Germany (6):
  - Kerckhoff-Klinik gGmbH, Bad Nauheim, Hesse
  - Rheumapraxis Dr. med. Reiner Kurthen, Aachen, North Rhine-Westphalia
  - Studienambulanz Dr. Wassenberg, Ratingen, North Rhine-Westphalia
  - SMO.MD GmbH, Magdeburg, Saxony-Anhalt
  - Klinische Forschung Berlin-Mitte GmbH, Berlin
  - HRF Hamburger Rheuma Forschungszentrum, Hamburg
- Hungary (8):
  - Principal SMO Kft., Baja
  - DRC Gyogyszervizsgalo Kozpont Kft., Balatonfüred
  - Clinexpert Kft., Budapest
  - Obudai Egeszsegugyi Centrum Kft., Budapest
  - Kiskunhalasi Semmelweis Korhaz, Kiskunhalas
  - DRC Szekesfehervar, Székesfehérvár
  - MAV Korhaz es Rendelointezet, Szolnok
  - Vital-Medicina Kft., Veszprém
- Dr.Saulite-Kandevica Private Practice, Liepāja, Latvia
- Lithuania (6):
  - Alytus Regional S. Kudirkos Hospital, Public Institution, Alytus
  - Republican Kaunas Hospital, Public Institution, Kaunas
  - Klaipeda University Hospital, Public Institution, Klaipėda
  - Siauliai Republican Hospital, Public Institution, Šiauliai
  - Center Outpatient Clinic, Public Institution, Vilnius
  - Vilnius University Hospital Santariskiu Clinics, Public Institution, Vilnius
- Mexico (11):
  - Clinica de Investigacion en Reumatologia y Obesidad S.C., Guadalajara, Jalisco
  - Centro de Estudios de Investigacion Basica y Clinica SC, Guadalajara, Jalisco
  - Clinicos Asociados BOCM S.C., Mexico City, Mexico City
  - Centro de Investigacion Clínica GRAMEL S.C, Mexico City, Mexico City
  - Comite Mexicano Para la Prevencion de Osteoporosis AC, Mexico City, Mexico City
  - Clinstile, S.A. de C.V., Mexico City, Mexico City
  - Accelerium S. de R.L. de C.V., Monterrey, Nuevo León
  - Universidad Autonoma de Nuevo Leon, Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Investigacion y Biomedicina de Chihuahua, S.C., Chihuahua City
  - Clinical Research Institute S.C., Mexico City
  - Centro de Alta Especialidad en Reumatología e Investigación del Potosí, S.C., San Luis Potosí City
- Poland (19):
  - CERMED, Bialystok
  - ZDROWIE Osteo-Medic, Bialystok
  - Szpital Uniwersytecki nr 2 im.dr J. Biziela, Bydgoszcz
  - MCBK Iwona Czajkowska Anna Podrażka- Szczepaniak S.C., Grodzisk Mazowiecki
  - Polimedica Centrum Badań, Profilaktyki I Leczenia, Kielce
  - CCBR - Lodz - PL, Lodz
  - Centrum Medyczne AMED, Lodz
  - ETYKA Osrodek Badan Klinicznych, Olsztyn
  - Szpital Wojewodzki im. Prymasa Kardynala Stefana Wyszynskiego, Sieradz
  - Clinmed Research, Skierniewice
  - RCMed, Sochaczew
  - KO-MED Centra Kliniczne Staszow, Staszów
  - Samodzielny Publiczny ZOZ Tomaszow Lubelski, Tomaszów Lubelski
  - Nasz lekarz Przychodnie Medyczne, Torun
  - Medycyna Kliniczna, Warsaw
  - Rheuma Medicus Zaklad Opieki Zdrowotnej, Warsaw
  - McM Polimedica, Warsaw
  - KO-MED Centra Kliniczne Zamosc, Zamość
  - Santa Familia Centrum Badan, Profilaktyki i Leczenia, Zgierz
- Russia (34):
  - FSBEI HE "Altai State Medical University of the Ministry of Healthcare of Russian Federation", Barnaul, Altayskiy Kray
  - SAHI of Kemerovo region "Regional Clinical Hospital for War Veterans", Kemerovo, Kemerovo Oblast
  - Medical Center LLC "Maksimum Zdoroviya", Kemerovo, Kemerovo Oblast
  - Budgetary Healthcare Institution "Kursk Regional Clinical Hospital" of Healthcare Committee of Kursk region, Kursk, Kursk Oblast
  - SPb SBHI "Clinical Rheumatological Hospital #25", Fourth Rheumatology Unit, Saint Petersburg, Leningradskaya Oblast'
  - SBHI of Moscow "City Clinical Hospital No.1 n.a. Pirogov" Healthcare Department of Moscow, Moscow, Moscovskaya Oblast
  - FSAEI HE "First MSMU n.a. I.M. Sechenov of the Ministry of Health of the Russian Federation" University Clinical Hospital No.1, Moscow, Moscovskaya Oblast
  - FSAEI HE "First MSMU n.a. I.M. Sechenov of the Ministry of Health of the Russian Federation", Moscow, Moscovskaya Oblast
  - State Budgetary Healthcare Institution "City Clinical Hospital # 15 n.a O.M. Filatov" of Moscow Healtheare Department, Moscow, Moscow Oblast
  - SBHI of Moscow "City Clinical Hospital #4 of Moscow Healthcare Departament", Moscow, Moscow Oblast
  - SBHI of Nizhegorodsky Region "State Clinical Hospital #5 of Nizhegorodsky District of Nizhny Novgorod", Nizhny Novgorod, Nizhny Novgorod Oblast
  - SBHI of Nizhny Novgorod Region "Nizhny Novgorod Regional Clinical Hospital n.a.Semashko", Nizhny Novgorod, Nizhny Novgorod Oblast
  - State Autonomous Healthcare Institution of Novosibirsk region "City Polyclinic #1", Novosibirsk, Novosibirsk Oblast
  - LLC "Clinical Diagnostic Center "Ultramed", Omsk, Omsk Oblast
  - Budgetary Healthcare Institution of Omsk Region "Regional Clinical Hospital", Omsk, Omsk Oblast
  - SBHI of the Republic of Karelia "Republican Hospital named after V.A. Baranov", Petrozavodsk, Republic of Karelia
  - State Budgetary Healthcare Institution "Republican Clinical Hospital n.a. G.G. Kuvatov", Ufa, Respublic of Bashkortostan
  - FSBEI HE "Rostov State Medical Unversity" of Ministry of Health of the Russian Federation, Rostov-on-Don, Rostov Oblast
  - FSBEI HE 'Ryazan State Medical University n.a. I.P.Pavlov" of the Ministry of Health of Russian Federation, Ryazan, Ryazan Oblast
  - FSBEI HE "Saratov SMU n.a. V.I.Razumovsky of Ministry of Health of Russian Federation", Saratov, Saratov Oblast
  - State Healthcare Institution "Regional Clinical Hospital", Saratov, Saratov Oblast
  - Private Healthcare Institution "Clinical Hospital Russian Railways-Medicine of City Smolensk", Smolensk, Smolensk Oblast
  - FSBEI HE StSMU MOH Russia based on SBHI of Stavropol Region "Stavropol Regional Clinical Hospital", Stavropol, Stavropol Kray
  - State Autonomous Healthcare Institution of Sverdlovsk Region "Sverdlovsk Regional Clinical Hospital No.1", Yekaterinburg, Sverdlovsk Oblast
  - FSBEI HE "Ural State Medical University" of Ministry of Health of Russian Federation based on MBI "Central City Clinical Hospital No.6", Yekaterinburg, Sverdlovsk Oblast
  - FSBEI HE "Kazan State Medical University of the Ministry of Health of the Russian Federation" on the base of SAHI "Republican Clinical Hospital of the Ministry of Health of Tatarstan Republic", Kazan', The Republic of Tatarstan
  - State Healthcare Institution of Tula region "Tula Regional Clinical Hospital", Tula, Tulskaya Oblast
  - State Healthcare Institution "Ulyanovsk Regional Clinical Hospital", Ulyanovsk, Ulyanovsk Oblast
  - SBHI of Vladimir Region "Regional Clinical Hospital", Rheumatology Departament, Vladimir, Vladimirskaya Oblast’
  - SBHI "Yaroslavl Regional Clinical Hospital", Rheumatology department, Yaroslavl, Yaroslavl Oblast
  - State Autonomous Helthcare Institution of Yaroslavl region "Clinical Hospital of Emergency Care n.a. Solovyev", Yaroslavl, Yaroslavsakaya Oblast
  - FSBSI "Scientific Research Institute of Rheumatology n.a. V.A. Nasonova", Moscow
  - FSAEI HE "First MSMU n.a. I.M. Sechenov of the Ministry of Health of the Russian Federation", Moscow
  - FSBI "National Medical Research Center n.a. V.A.Almazov" of the Ministry of Healthcare of the Russian Federation, Saint Petersburg
- South Korea (7):
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Eulji University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Jeju National University Hospital, Jeju City
  - Severance Hospital, Yonsei University No. 31 Office, Pediatric Oncology Clinic, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Taiwan (2):
  - Chi Mei Medical Center, Yung Kang Branch, Tainan
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District
- United Kingdom (6):
  - Torbay Hospital, Torquay, Devon
  - Whipps Cross University Hospital, London, Greater London
  - Royal Free Hospital, London, Greater London
  - Basingstoke and North Hampshire Hospital, Basingstoke, Hampshire
  - Maidstone Hospital, Maidstone, Kent
  - Arrowe Park Hospital, Metropolitan Borough of Wirral, Merseyside

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was conducted at 241 sites in 18 countries (Argentina, Belarus, Bulgaria, Brazil, Colombia, Czech Republic, Germany, Estonia, United Kingdom, Hungary, South Korea, Lithuania, Latvia, Mexico, Poland, Russia, Taiwan, United States).
  A total of 2105 subjects who had previously completed 24 weeks of double-blind treatment in a core study were randomized. All except one randomized subject received OKZ treatment. A total of 2104 subjects were analyzed for efficacy in the mITT Population.
Groups:
- Treatment Arm 1: OKZ 64 mg q4w + MTX: Olokizumab 64 mg subcutaneous (SC) q4w + concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular).
  Olokizumab 64 mg SC q4w: 160 mg/mL sterile solution for SC injection in a 2 mL clear Type I glass vial with target volume of 0.4 mL or in the pre-filled syringe (PFS). PFS is composed of a 1 mL clear Type I glass barrel vial with target volume of 0.4 mL.
Period: Overall Study
Arm/Group | Treatment Arm 1: OKZ 64 mg q4w + MTX | Treatment Arm 2: OKZ 64 mg q2w + MTX
Started | 1058 (One subject was randomized in error and did not receive any dose of study drug.) | 1047
mITT | 1057 | 1047
Safety Population | 1043 (Subjects in the safety population were analyzed according to the treatment they actually received during the OLE study. (14 patients had been assigned to q4w group but actually received the treatment according to the q2w group).) | 1061 (Subjects in the safety population were analyzed according to the treatment they actually received during the OLE study. (14 patients had been assigned to q4w group but actually received the treatment according to the q2w group).)
Completed | 830 | 844
Not Completed | 228 | 203
Not completed — randomized in error | 1 | 0
Not completed — Death | 13 | 13
Not completed — Lost to Follow-up | 23 | 13
Not completed — Withdrawal by Subject | 139 | 124
Not completed — Covid-19 | 43 | 34
Not completed — Patient Moved Out Of Residence And was Not Able To Come To The Site | 1 | 3
Not completed — Lack Of Discipline In Adhering To The Schedule Of Visits, Difficult Cooperation With The Patient | 1 | 0
Not completed — Safety Follow-Up Visit (SFU)-3 Was Performed By Phone Due To Family Reasons | 1 | 0
Not completed — Patient Completed The Treatment, But Could Not Come For Follow-Up Visits Due To Another City Moving | 1 | 0
Not completed — Site was closed | 2 | 3
Not completed — Study Coordinator Error, Patient Started A Biologic And Study Coordinator Forgot To Complete SFU | 1 | 0
Not completed — Principal Investigator (PI) Decision, The PI Starting Subject On Another Biologic Medication | 0 | 1
Not completed — PI Terminated Subject From IP (Ae's Abnormal Wbc, Abnormal Absolute Neutrophils Lab) | 1 | 0
Not completed — Patient Was Hospitalized Due To The SAE And Couldn't Visit The Site For Sfu-3 | 1 | 0
Not completed — Other: Adverse Event | 0 | 1
Not completed — Due To The Death Of His Wife, He Refused To Participate In Follow Up 3 | 0 | 1
Not completed — Follow Up Visit Not Performed (Patient Outside Residence) | 0 | 2
Not completed — Subject Refusal To Attend Visit | 0 | 1
Not completed — Personal Reasons | 0 | 1
Not completed — PI Did Not Feel It Was Best For Subject To Be Without Treatment For 12 Weeks. | 0 | 1
Not completed — Lack Of Efficacy (PI Perspective) End Of Study Visit | 0 | 1
Not completed — Compliance With Medication | 0 | 1
Not completed — Subject Has A Severe Or Life Threatening Infection That Requires Hospitalization Per Medical Monitor | 0 | 1
Not completed — Other: Protocol Violation (Refused From SFU Visits) | 0 | 1
Not completed — Study Terminated By Principal Investigator | 0 | 1

BASELINE CHARACTERISTICS:
Population: Subjects who received OKZ in the core study received the same OKZ treatment regimen in the OLE study. Subjects who received in the core study placebo or adalimumab were randomized 1:1 to OKZ 64 mg q2w or OKZ 64 mg q4w regimens in the OLE study. The mITT population included all subjects who signed an ICF for participation in the OLE study, were randomized in the OLE study, received at least 1 dose of study treatment in the OLE study (1057 subjects (OKZ 64 mg q4w), 1047 subjects (OKZ 64 mg q2w)).
Groups:
- Treatment Arm 1: OKZ 64 mg q4w + MTX: Olokizumab 64 mg SC q4w + concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular).
  Olokizumab 64 mg SC q4w: 160 mg/mL sterile solution for SC injection in a 2 mL clear Type I glass vial with target volume of 0.4 mL or in the pre-filled syringe (PFS). PFS is composed of a 1 mL clear Type I glass barrel vial with target volume of 0.4 mL.
- Total: Total of all reporting groups
Arm/Group | Treatment Arm 1: OKZ 64 mg q4w + MTX | Treatment Arm 2: OKZ 64 mg q2w + MTX | Total
Number analyzed (Participants) | 1057 | 1047 | 2104
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (12.05) | 53.7 (11.78) | 53.7 (11.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 851 | 840 | 1691
  Male | 206 | 207 | 413
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 357 | 332 | 689
  Not Hispanic or Latino | 700 | 715 | 1415
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 15 | 17 | 32
  Black or African American | 31 | 46 | 77
  White | 914 | 896 | 1810
  Other/Mixed | 97 | 88 | 185
Region of Enrollment [Count of Participants; unit: Participants]
  Colombia | 32 | 32 | 64
  Argentina | 81 | 73 | 154
  Hungary | 31 | 36 | 67
  United States | 150 | 155 | 305
  Czechia | 105 | 94 | 199
  United Kingdom | 3 | 6 | 9
  Belarus | 9 | 9 | 18
  Russia | 217 | 208 | 425
  Latvia | 1 | 2 | 3
  South Korea | 6 | 6 | 12
  Taiwan | 4 | 4 | 8
  Brazil | 55 | 61 | 116
  Poland | 138 | 133 | 271
  Mexico | 137 | 127 | 264
  Bulgaria | 36 | 41 | 77
  Lithuania | 29 | 38 | 67
  Germany | 16 | 20 | 36
  Estonia | 7 | 2 | 9
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 28.201 [14.88 to 56.25] | 28.229 [15.62 to 62.22] | 28.215 [14.88 to 62.22]

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events (AEs), by System Organ Class and Preferred Term (Safety Population)
Description: Incidence of Treatment-Emergent Adverse Events Reported for ≥5% of Subjects in Any Treatment Group by System Organ Class or Preferred Term
Time Frame: up to Week 126
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm 1: OKZ 64 mg q4w + MTX | Treatment Arm 2: OKZ 64 mg q2w + MTX
Number analyzed (Participants) | 1043 | 1061
Participants
  Infections and infestations | 401 | 408
  Infections and infestations: Nasopharyngitis | 71 | 87
  Infections and infestations: Upper respiratory tract infection | 59 | 67
  Infections and infestations: Bronchitis | 59 | 45
  Investigations | 284 | 290
  Investigations: Alanine aminotransferase increased | 97 | 118
  Investigations: Aspartate aminotransferase increased | 52 | 63
  Musculoskeletal and connective tissue disorders | 149 | 152
  Blood and lymphatic system disorders | 125 | 147
  Blood and lymphatic system disorders: Leukopenia | 46 | 60
  Blood and lymphatic system disorders: Neutropenia | 42 | 57
  Metabolism and nutrition disorders | 113 | 135
  Gastrointestinal disorders | 100 | 118
  Injury, poisoning and procedural complications | 101 | 95
  Skin and subcutaneous tissue disorders | 88 | 94
  Nervous system disorders | 60 | 81
  Respiratory, thoracic and mediastinal disorders | 60 | 68
  Vascular disorders | 60 | 68
  General disorders and administration site conditions | 54 | 65

2. Primary Outcome: Incidence of Treatment-Emergent Serious Adverse Events (SAEs), by System Organ Class and Preferred Term (Safety Population)
Description: Incidence of Serious Treatment-Emergent Adverse Events by System Organ Class or Preferred Term.
  Deaths are included.
Time Frame: up to Week 126
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm 1: OKZ 64 mg q4w + MTX | Treatment Arm 2: OKZ 64 mg q2w + MTX
Number analyzed (Participants) | 1043 | 1061
Participants
  Number of Subjects with at Least One SAE | 129 | 120
  Infections and infestations | 40 | 47
  Infections and infestations: Pneumonia | 7 | 7
  Infections and infestations: Cellulitis | 7 | 4
  Infections and infestations: Erysipelas | 5 | 4
  Infections and infestations: COVID-19 | 1 | 3
  Infections and infestations: Pyelonephritis acute | 2 | 2
  Infections and infestations: COVID-19 pneumonia | 2 | 1
  Infections and infestations: Pyelonephritis | 2 | 1
  Infections and infestations: Sepsis | 0 | 3
  Infections and infestations: Abscess limb | 1 | 1
  Infections and infestations: Diverticulitis | 1 | 1
  Infections and infestations: Osteomyelitis | 1 | 1
  Infections and infestations: Abdominal wall abscess | 0 | 1
  Infections and infestations: Abscess soft tissue | 0 | 1
  Infections and infestations: Acute sinusitis | 0 | 1
  Infections and infestations: Atypical pneumonia | 1 | 0
  Infections and infestations: Bartholinitis | 0 | 1
  Infections and infestations: Bronchitis | 0 | 1
  Infections and infestations: Bullous erysipelas | 1 | 0
  Infections and infestations: Bursitis infective | 0 | 1
  Infections and infestations: Cat scratch disease | 0 | 1
  Infections and infestations: Dengue fever | 0 | 1
  Infections and infestations: Device related infection | 0 | 1
  Infections and infestations: Device related sepsis | 0 | 1
  Infections and infestations: Encephalomyelitis | 0 | 1
  Infections and infestations: Gangrene | 0 | 1
  Infections and infestations: Gastroenteritis | 0 | 1
  Infections and infestations: Influenza | 0 | 1
  Infections and infestations: Intervertebral discitis | 1 | 0
  Infections and infestations: Joint abscess | 1 | 0
  Infections and infestations: Latent tuberculosis | 0 | 1
  Infections and infestations: Localised infection | 1 | 0
  Infections and infestations: Lower respiratory tract infection | 0 | 1
  Infections and infestations: Ludwig angina | 1 | 0
  Infections and infestations: Medical device site abscess | 0 | 1
  Infections and infestations: Necrotising fasciitis | 0 | 1
  Infections and infestations: Necrotising soft tissue infection | 0 | 1
  Infections and infestations: Post procedural infection | 1 | 0
  Infections and infestations: Pulmonary tuberculosis | 0 | 1
  Infections and infestations: Renal abscess | 1 | 0
  Infections and infestations: Salpingo-oophoritis | 1 | 0
  Infections and infestations: Scrotal abscess | 1 | 0
  Infections and infestations: Septic shock | 0 | 1
  Infections and infestations: Streptococcal sepsis | 1 | 0
  Infections and infestations: Tonsillitis | 0 | 1
  Infections and infestations: Urinary tract infection | 0 | 1
  Infections and infestations: Viral infection | 0 | 1
  Infections and infestations: Viral upper respiratory tract infection | 1 | 0
  Infections and infestations: Wound infection pseudomonas | 1 | 0
  Musculoskeletal and connective tissue disorders | 14 | 11
  Musculoskeletal and connective tissue disorders: Osteoarthritis | 6 | 6
  Musculoskeletal and connective tissue disorders: Osteonecrosis | 1 | 1
  Musculoskeletal and connective tissue disorders: Rheumatoid arthritis | 1 | 1
  Musculoskeletal and connective tissue disorders: Arthritis | 1 | 0
  Musculoskeletal and connective tissue disorders: Bursitis | 1 | 0
  Musculoskeletal and connective tissue disorders: Cervical spinal stenosis | 0 | 1
  Musculoskeletal and connective tissue disorders: Foot deformity | 0 | 1
  Musculoskeletal and connective tissue disorders: Intervertebral disc protrusion | 1 | 0
  Musculoskeletal and connective tissue disorders: Joint ankylosis | 0 | 1
  Musculoskeletal and connective tissue disorders: Muscle contracture | 1 | 0
  Musculoskeletal and connective tissue disorders: Musculoskeletal chest pain | 1 | 0
  Musculoskeletal and connective tissue disorders: Spinal osteoarthritis | 1 | 0
  Injury, poisoning and procedural complications | 8 | 14
  Injury, poisoning and procedural complications: Clavicle fracture | 1 | 1
  Injury, poisoning and procedural complications: Femoral neck fracture | 0 | 2
  Injury, poisoning and procedural complications: Head injury | 2 | 0
  Injury, poisoning and procedural complications: Hip fracture | 0 | 2
  Injury, poisoning and procedural complications: Acetabulum fracture | 0 | 1
  Injury, poisoning and procedural complications: Arthropod bite | 1 | 0
  Injury, poisoning and procedural complications: Comminuted fracture | 0 | 1
  Injury, poisoning and procedural complications: Concussion | 0 | 1
  Injury, poisoning and procedural complications: Extradural haematoma | 1 | 0
  Injury, poisoning and procedural complications: Femur fracture | 1 | 0
  Injury, poisoning and procedural complications: Foot fracture | 0 | 1
  Injury, poisoning and procedural complications: Humerus fracture | 0 | 1
  Injury, poisoning and procedural complications: Lower limb fracture | 0 | 1
  Injury, poisoning and procedural complications: Multiple injuries | 1 | 0
  Injury, poisoning and procedural complications: Muscle rupture | 1 | 0
  Injury, poisoning and procedural complications: Overdose | 0 | 1
  Injury, poisoning and procedural complications: Post procedural complication | 0 | 1
  Injury, poisoning and procedural complications: Thoracic vertebral fracture | 0 | 1
  Injury, poisoning and procedural complications: Traumatic intracranial haematoma | 0 | 1
  Injury, poisoning and procedural complications: Wrist fracture | 0 | 1
  Cardiac disorders | 11 | 10
  Cardiac disorders: Acute myocardial infarction | 3 | 0
  Cardiac disorders: Arrhythmia | 1 | 1
  Cardiac disorders: Atrial fibrillation | 0 | 2
  Cardiac disorders: Acute coronary syndrome | 0 | 1
  Cardiac disorders: Angina unstable | 1 | 0
  Cardiac disorders: Atrioventricular block complete | 1 | 0
  Cardiac disorders: Atrioventricular block second degree | 1 | 0
  Cardiac disorders: Bradycardia | 0 | 1
  Cardiac disorders: Cardiac arrest | 1 | 0
  Cardiac disorders: Cardiac failure chronic | 0 | 1
  Cardiac disorders: Cardiac failure congestive | 0 | 1
  Cardiac disorders: Coronary artery occlusion | 1 | 0
  Cardiac disorders: Coronary artery stenosis | 0 | 1
  Cardiac disorders: Myocardial infarction | 0 | 1
  Cardiac disorders: Right ventricular dysfunction | 0 | 1
  Cardiac disorders: Sinus tachycardia | 0 | 1
  Cardiac disorders: Stress cardiomyopathy | 1 | 0
  Cardiac disorders: Supraventricular tachyarrhythmia | 0 | 1
  Cardiac disorders: Ventricular fibrillation | 1 | 0
  Gastrointestinal disorders | 8 | 12
  Gastrointestinal disorders: Diverticular perforation | 1 | 2
  Gastrointestinal disorders: Abdominal pain | 1 | 1
  Gastrointestinal disorders: Colitis | 1 | 1
  Gastrointestinal disorders: Gastritis erosive | 0 | 2
  Gastrointestinal disorders: Abdominal hernia obstructive | 1 | 0
  Gastrointestinal disorders: Dyspepsia | 0 | 1
  Gastrointestinal disorders: Gastric polyps | 1 | 0
  Gastrointestinal disorders: Gastric ulcer | 0 | 1
  Gastrointestinal disorders: Gastrointestinal disorder | 0 | 1
  Gastrointestinal disorders: Intestinal obstruction | 0 | 1
  Gastrointestinal disorders: Obstructive pancreatitis | 1 | 0
  Gastrointestinal disorders: Pancreatitis acute | 0 | 1
  Gastrointestinal disorders: Pancreatitis chronic | 1 | 0
  Gastrointestinal disorders: Peptic ulcer | 1 | 0
  Gastrointestinal disorders: Salivary gland calculus | 0 | 1
  Neoplasms benign, malignant and unspecified (incl cysts and polyps) | 11 | 8
  Neoplasms benign, malignant and unspecified: Meningioma | 1 | 1
  Neoplasms benign, malignant and unspecified: Benign neoplasm of thyroid gland | 1 | 0
  Neoplasms benign, malignant and unspecified: Central nervous system neoplasm | 0 | 1
  Neoplasms benign, malignant and unspecified: Cervix carcinoma stage II | 1 | 0
  Neoplasms benign, malignant and unspecified: Clear cell renal cell carcinoma | 1 | 0
  Neoplasms benign, malignant and unspecified: Colon cancer | 1 | 0
  Neoplasms benign, malignant and unspecified: Endometrial adenocarcinoma | 1 | 0
  Neoplasms benign, malignant and unspecified: Endometrial cancer | 0 | 1
  Neoplasms benign, malignant and unspecified: Extranodal marginal zone B-cell lymphoma (MALT type) | 0 | 1
  Neoplasms benign, malignant and unspecified: Gastric cancer | 1 | 0
  Neoplasms benign, malignant and unspecified: Invasive ductal breast carcinoma | 0 | 1
  Neoplasms benign, malignant and unspecified: Lung adenocarcinoma stage III | 1 | 0
  Neoplasms benign, malignant and unspecified: Malignant melanoma | 1 | 0
  Neoplasms benign, malignant and unspecified: Marginal zone lymphoma | 0 | 1
  Neoplasms benign, malignant and unspecified: Meningioma benign | 1 | 0
  Neoplasms benign, malignant and unspecified: Metastatic neoplasm | 1 | 0
  Neoplasms benign, malignant and unspecified: Pancreatic carcinoma metastatic | 0 | 1
  Neoplasms benign, malignant and unspecified: Salivary gland cancer | 1 | 0
  Neoplasms benign, malignant and unspecified: Uterine leiomyoma | 0 | 1
  Nervous system disorders | 13 | 6
  Nervous system disorders: Cerebrovascular accident | 4 | 2
  Nervous system disorders: Dizziness | 1 | 1
  Nervous system disorders: Ischaemic stroke | 0 | 2
  Nervous system disorders: Syncope | 2 | 0
  Nervous system disorders: Carotid artery aneurysm | 1 | 0
  Nervous system disorders: Encephalopathy | 1 | 0
  Nervous system disorders: Migraine | 1 | 0
  Nervous system disorders: Myelopathy | 1 | 0
  Nervous system disorders: Paraesthesia | 1 | 0
  Nervous system disorders: Pineal gland cyst | 1 | 0
  Nervous system disorders: Seizure | 1 | 0
  Nervous system disorders: Subarachnoid haemorrhage | 0 | 1
  Nervous system disorders: Transient ischaemic attack | 1 | 0
  Respiratory, thoracic and mediastinal disorders | 7 | 12
  Respiratory, thoracic and mediastinal disorders: Pulmonary embolism | 2 | 4
  Respiratory, thoracic and mediastinal disorders: Chronic obstructive pulmonary disease | 1 | 1
  Respiratory, thoracic and mediastinal disorders: Pulmonary fibrosis | 1 | 1
  Respiratory, thoracic and mediastinal disorders: Respiratory failure | 1 | 1
  Respiratory, thoracic and mediastinal disorders: Asthmatic crisis | 1 | 0
  Respiratory, thoracic and mediastinal disorders: Bronchitis chronic | 0 | 1
  Respiratory, thoracic and mediastinal disorders: Chronic respiratory failure | 0 | 1
  Respiratory, thoracic and mediastinal disorders: Chylothorax | 0 | 1
  Respiratory, thoracic and mediastinal disorders: effusion | 1 | 0
  Respiratory, thoracic and mediastinal disorders: Pleurisy | 0 | 1
  Respiratory, thoracic and mediastinal disorders: Pneumothorax | 0 | 1
  Investigations | 9 | 6
  Investigations: Alanine aminotransferase increased | 7 | 5
  Investigations: Hepatic enzyme increased | 1 | 1
  Investigations: Liver function test increased | 1 | 0
  Hepatobiliary disorders | 6 | 3
  Hepatobiliary disorders: Cholelithiasis | 2 | 1
  Hepatobiliary disorders: Cholecystitis chronic | 1 | 1
  Hepatobiliary disorders: Biliary colic | 1 | 0
  Hepatobiliary disorders: Hepatotoxicity | 1 | 0
  Hepatobiliary disorders: Hyperplastic cholecystopathy | 0 | 1
  Hepatobiliary disorders: Liver injury | 1 | 0
  General disorders and administration site conditions | 4 | 4
  General disorders and administration site conditions: Death | 1 | 1
  General disorders and administration site conditions: Sudden death | 1 | 1
  General disorders and administration site conditions: Lithiasis | 1 | 0
  General disorders and administration site conditions: Pyrexia | 0 | 1
  General disorders and administration site conditions: Sudden cardiac death | 1 | 0
  General disorders and administration site conditions: Vascular stent occlusion | 0 | 1
  Reproductive system and breast disorders | 3 | 3
  Reproductive system and breast disorders: Uterine polyp | 2 | 0
  Reproductive system and breast disorders: Endometrial hyperplasia | 0 | 1
  Reproductive system and breast disorders: Female genital tract fistula | 0 | 1
  Reproductive system and breast disorders: Genital haemorrhage | 1 | 0
  Reproductive system and breast disorders: Intermenstrual bleeding | 0 | 1
  Reproductive system and breast disorders: Ovarian cyst | 0 | 1
  Skin and subcutaneous tissue disorders | 4 | 2
  Skin and subcutaneous tissue disorders: Dermatitis | 1 | 1
  Skin and subcutaneous tissue disorders: Skin ulcer | 1 | 1
  Skin and subcutaneous tissue disorders: Dermatitis contact | 1 | 0
  Skin and subcutaneous tissue disorders: Erythema | 1 | 0
  Vascular disorders | 4 | 2
  Vascular disorders: Deep vein thrombosis | 1 | 0
  Vascular disorders: Hypertensive crisis | 1 | 0
  Vascular disorders: Peripheral artery occlusion | 0 | 1
  Vascular disorders: Shock haemorrhagic | 1 | 0
  Vascular disorders: Thrombophlebitis | 0 | 1
  Vascular disorders: Varicose vein | 1 | 0
  Renal and urinary disorders | 3 | 2
  Renal and urinary disorders: Calculus urinary | 1 | 0
  Renal and urinary disorders: Nephritis | 1 | 0
  Renal and urinary disorders: Nephrolithiasis | 0 | 1
  Renal and urinary disorders: Renal colic | 1 | 0
  Renal and urinary disorders: Ureterolithiasis | 0 | 1
  Blood and lymphatic system disorders | 1 | 2
  Blood and lymphatic system disorders: Febrile neutropenia | 0 | 1
  Blood and lymphatic system disorders: Lymphadenopathy | 1 | 0
  Blood and lymphatic system disorders: Splenic cyst | 0 | 1
  Pregnancy, puerperium and perinatal conditions | 2 | 1
  Pregnancy, puerperium and perinatal conditions: Abortion spontaneous | 1 | 0
  Pregnancy, puerperium and perinatal conditions: Abortion threatened | 1 | 0
  Pregnancy, puerperium and perinatal conditions: Ectopic pregnancy | 0 | 1
  Ear and labyrinth disorders | 1 | 1
  Ear and labyrinth disorders: Deafness neurosensory | 0 | 1
  Ear and labyrinth disorders: Vestibular disorder | 1 | 0
  Eye disorders | 0 | 2
  Eye disorders: Cataract | 0 | 1
  Eye disorders: Ocular myasthenia | 0 | 1
  Immune system disorders | 1 | 0
  Immune system disorders: Hypersensitivity | 1 | 0
  Psychiatric disorders | 1 | 0
  Psychiatric disorders: Completed suicide | 1 | 0

3. Primary Outcome: Incidence of Treatment-Emergent Adverse Events of Special Interest (AESI)
Time Frame: up to Week 126
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Arm 1: OKZ 64 mg q4w + MTX: Olokizumab 64 mg SC q4w + concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular).
  Olokizumab 64 mg SC q4w: 160 mg/mL sterile solution for SC injection in a 2 mL clear Type I glass vial with target volume of 0.4 mL or in the pre-filled syringe (PFS).PFS is composed of a 1 mL clear Type I glass barrel vial with target volume of 0.4 mL.
  Concomitant treatment: Methotrexate 15 to 25 mg/week (or ≥ 10 mg/week if there was documented intolerance to higher doses). (Subject maintained their stable dose and route (oral, SC, or IM) during the core study and for ≥ 12 additional weeks of OLE.)
  Folic acid ≥ 5 mg per week or equivalent
- Treatment Arm 2: OKZ 64 mg q2w + MTX: Olokizumab 64 mg SC q2w + concomitant background therapy (Methotrexate) at a stable dose with a stable route of administration (oral, subcutaneous, or intramuscular).
  Olokizumab 64 mg SC q2w: 160 mg/mL sterile solution for SC injection in a 2 mL clear Type I glass vial with target volume of 0.4 mL or in the pre-filled syringe (PFS). PFS is composed of a 1 mL clear Type I glass barrel vial with target volume of 0.4 mL.
  Concomitant treatment: Methotrexate 15 to 25 mg/week (or ≥ 10 mg/week if there was documented intolerance to higher doses). (Subject maintained their stable dose and route (oral, SC, or IM) during the core study and for ≥ 12 additional weeks of OLE.)
  Folic acid ≥ 5 mg per week or equivalent
Arm/Group | Treatment Arm 1: OKZ 64 mg q4w + MTX | Treatment Arm 2: OKZ 64 mg q2w + MTX
Number analyzed (Participants) | 1043 | 1061
Participants
  Infections | 389 | 398
  Infections: Opportunistic Infections | 19 | 22
  Malignancies | 9 | 6
  Basal cell carcinoma | 2 | 1
  Elevation of Blood Lipids | 120 | 138
  Systemic Injection Reactions and Hypersensitivity Reactions | 99 | 100
  Systemic Injection Reactions and Hypersensitivity Reactions: Anaphylactic Reactions | 0 | 0
  Gastrointestinal Perforations | 1 | 2
  Neutropenia, Thrombocytopenia, Leukocytopenia and Pancytopenia | 146 | 168
  Potential Hepatotoxicity | 68 | 63
  Injection Site Reactions | 34 | 34
  Demyelination in Peripheral or Central Nervous System | 0 | 1
  Autoimmune Disorders | 48 | 41

4. Primary Outcome: Incidence of Treatment-Emergent AEs Leading to Withdrawal of the Study Treatment
Time Frame: up to Week 126
Population: Safety Population (3 Subjects discontinued treatment due to an AE but they did not have an AE that led to treatment discontinuation.)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm 1: OKZ 64 mg q4w + MTX | Treatment Arm 2: OKZ 64 mg q2w + MTX
Number analyzed (Participants) | 1043 | 1061
Participants | 87 | 90

5. Primary Outcome: Incidence Rate of Treatment Emergent AEs Per Patient-years of Exposure
Description: Incidence Rate of all Subjects with at Least One Treatment Emergent AE. Subject Incidence Rate (IR) is summarized per 100 subject years (SY) of follow-up (/100 SY) based on the OLE safety population and presented by study treatments.
Time Frame: up to Week 126
Measure: Number; unit: subjects per 100 subject-years
Groups:
- OKZ 64 mg q4w: subjects receiving OKZ 64 mg q4w during the core study or OLE
- OKZ 64 mg q2w: subjects receiving OKZ 64 mg q2w during the core study or OLE
Arm/Group | OKZ 64 mg q4w | OKZ 64 mg q2w
Number analyzed (Participants) | 1043 | 1061
subjects per 100 subject-years | 48.75 | 49.84

6. Primary Outcome: Incidence Rate of Treatment Emergent SAEs Per Patient-years of Exposure
Description: Incidence Rate of all Subjects with at Least One Treatment Emergent SAE. Subject Incidence Rate (IR) is summarized per 100 subject years (SY) of follow-up (/100 SY) based on the OLE safety population and presented by study treatments.
Time Frame: up to Week 126
Measure: Number; unit: subjects per 100 subject-years
Arm/Group | OKZ 64 mg q4w | OKZ 64 mg q2w
Number analyzed (Participants) | 1043 | 1061
subjects per 100 subject-years | 7.74 | 7.37

7. Primary Outcome: Incidence Rate of Treatment Emergent AESIs (Safety Population)
Description: Incidence Rate of all Subjects with at Least One Treatment Emergent AESI. Subject Incidence Rate (IR) is summarized per 100 subject years (SY) of follow-up (/100 SY) based on the OLE safety population and presented by study treatments.
Time Frame: up to Week 126
Population: An AE is defined as treatment-emergent under a given study treatment, if AE's onset date is on or after the date of first dose the corresponding treatment and prior to initiation of the next study treatment, if any.
Measure: Number; unit: subjects per 100 subject-years
Arm/Group | OKZ 64 mg q4w | OKZ 64 mg q2w
Number analyzed (Participants) | 1043 | 1061
subjects per 100 subject-years | 40.49 | 42.13

8. Secondary Outcome: American College of Rheumatology 20% (ACR20) Response Rates Compare Against Core Baseline Through Week 82
Description: Number and Proportion of subjects achieving an ACR20 response who remain on randomized open-label treatment and in the study, assessed at several timepoints up to Week 82.
  American College of Rheumatology 20 % response is a composite defined as a ≥ 20% improvement from baseline in the swollen joint counts assessed in 66 joints and in the tender joint count assessed in 68 joints; and a ≥20% improvement from baseline in at least 3 of the 5 remaining core set measures:
  * Patient Global Assessment of Disease Activity (VAS)
  * Patient Assessment of Pain (VAS)
  * HAQ-DI
  * Physician Global Assessment (VAS)
  * Level of acute phase reactant (CRP)
Time Frame: up to Week 82
Population: mITT Population Intermediate missing data are imputed using surrounding visits. Response is calculated relative to the core baseline, the last available assessment prior to the first dose of the study treatment in the core study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm 1: OKZ 64 mg q4w + MTX | Treatment Arm 2: OKZ 64 mg q2w + MTX
Number analyzed (Participants) | 1057 | 1047
Participants
  Week 12 OLE | 861 | 863
  Week 20 OLE | 850 | 851
  Week 28 OLE | 839 | 829
  Week 40 OLE | 795 | 795
  Week 52 OLE | 780 | 783
  Week 64 OLE | 777 | 774
  Week 82 OLE | 811 | 830

9. Secondary Outcome: American College of Rheumatology 50% (ACR50) Response Rates Compare Against Core Baseline Through Week 82
Description: Number and Proportion of subjects achieving an ACR50 response who remain on randomized open-label treatment and in the study, assessed at several timepoints up to Week 82
  American College of Rheumatology 50 % response is a composite defined as a ≥ 50% improvement from baseline in the swollen joint counts assessed in 66 joints and in the tender joint count assessed in 68 joints; and a ≥ 50% improvement from baseline in at least 3 of the 5 remaining core set measures:
  * Patient Global Assessment of Disease Activity (VAS)
  * Patient Assessment of Pain (VAS)
  * HAQ-DI
  * Physician Global Assessment (VAS)
  * Level of acute phase reactant (CRP)
Time Frame: up to Week 82
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm 1: OKZ 64 mg q4w + MTX | Treatment Arm 2: OKZ 64 mg q2w + MTX
Number analyzed (Participants) | 1057 | 1047
Participants
  Week 12 OLE | 598 | 601
  Week 20 OLE | 607 | 607
  Week 28 OLE | 597 | 610
  Week 40 OLE | 600 | 594
  Week 52 OLE | 563 | 606
  Week 64 OLE | 584 | 583
  Week 82 OLE | 608 | 619

10. Secondary Outcome: American College of Rheumatology 70% (ACR70) Response Rates Compare Against Core Baseline Through Week 82
Description: Number and Proportion of subjects achieving an ACR70 response who remain on randomized open-label treatment and in the study, assessed at several timepoints up to Week 82
  American College of Rheumatology 70 % response is a composite defined as a ≥ 70% improvement from baseline in the swollen joint counts assessed in 66 joints and in the tender joint count assessed in 68 joints; and a ≥ 70% improvement from baseline in at least 3 of the 5 remaining core set measures:
  * Patient Global Assessment of Disease Activity (VAS)
  * Patient Assessment of Pain (VAS)
  * HAQ-DI
  * Physician Global Assessment (VAS)
  * Level of acute phase reactant (CRP)
Time Frame: up to Week 82
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm 1: OKZ 64 mg q4w + MTX | Treatment Arm 2: OKZ 64 mg q2w + MTX
Number analyzed (Participants) | 1057 | 1047
Participants
  Week 12 OLE | 330 | 362
  Week 20 OLE | 358 | 353
  Week 28 OLE | 367 | 357
  Week 40 OLE | 375 | 369
  Week 52 OLE | 370 | 387
  Week 64 OLE | 373 | 387
  Week 82 OLE | 382 | 393

11. Secondary Outcome: Proportion of Subjects With Simplified Disease Activity Index (SDAI) Remission Through Week 82
Description: The number and proportion of subjects with SDAI score ≤ 3.3 (considered to be in remission).
  The SDAI was calculated in the statistical database for analysis purposes using the SJC (28 joints), TJC (28 joints), CRP (mg/dL), the Patient Global Assessment of Disease Activity (VAS) (in cm), and the Physician Global Assessment (VAS) (in cm) according to the following formula: SJC + TJC + Patient Global Assessment of Disease Activity (VAS) + Physician Global Assessment (VAS) + CRP (mg/dL)
Time Frame: up to week 82
Population: Intermediate missing data are imputed using surrounding visits. The Core Baseline value was defined as the baseline value from the core study for subjects that enrol into the OLE study.The OLE Baseline value was defined as the last available measurement prior to the first OLE dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm 1: OKZ 64 mg q4w + MTX | Treatment Arm 2: OKZ 64 mg q2w + MTX
Number analyzed (Participants) | 1057 | 1047
Participants
  Core Baseline: number analyzed (Participants) | 1014 | 995
  Core Baseline | 0 | 0
  OLE Baseline: number analyzed (Participants) | 1057 | 1046
  OLE Baseline | 137 | 145
  Week 12 OLE | 161 | 190
  Week 20 OLE | 192 | 197
  Week 28 OLE | 196 | 196
  Week 40 OLE | 204 | 211
  Week 52 OLE | 218 | 225
  Week 64 OLE | 223 | 257
  Week 82 OLE | 231 | 267

12. Secondary Outcome: Disease Activity Score 28-joint Count (DAS28) Response Rates Through Week 82
Description: Number and Proportion of subjects with DAS28 low disease activity (based on DAS28 C-reactive protein (CRP) < 3.2), who remain on randomized open-label treatment and in the study, assessed at several timepoints up to Week 82.
  The DAS28 (CRP) was calculated in the statistical database for analysis purposes using the Swollen joint count (SJC) (28 joints), Tender joint count (TJC) (28 joints), CRP level, and the Patient Global Assessment of Disease Activity Visual Analog Scale (VAS) (100 mm VAS, where 0 is "no disease activity" and 100 was "maximal disease activity") according to the following formula: [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.36 × natural log (CRP+1)] + [0.014 × VAS] + 0.96.
Time Frame: up to Week 82
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm 1: OKZ 64 mg q4w + MTX | Treatment Arm 2: OKZ 64 mg q2w + MTX
Number analyzed (Participants) | 1057 | 1047
Participants
  Core Baseline: number analyzed (Participants) | 1044 | 1024
  Core Baseline | 1 | 1
  OLE Baseline: number analyzed (Participants) | 1057 | 1046
  OLE Baseline | 573 | 537
  Week 12 OLE | 681 | 685
  Week 20 OLE | 703 | 714
  Week 28 OLE | 684 | 694
  Week 40 OLE | 688 | 691
  Week 52 OLE | 679 | 680
  Week 64 OLE | 681 | 678
  Week 82 OLE | 706 | 712

13. Secondary Outcome: Change in Health Assessment Questionnaire-Disability Index (HAQ-DI) From Core Baseline at Week 12
Description: HAQ-DI Range: 0 (the best outcome) - 3 (the worst outcome), with a decrease from baseline indicating improvement.
  The HAQ-DI assesses the degree of difficulty experienced in 8 domains of daily living activities using 20 questions. The domains are dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities, and each domain (activity) consists of 2 or 3 items. For each question, the level of difficulty is scored from 0 to 3, where 0 = without any difficulty (the best outcome), 1 = with some difficulty, 2 = much difficulty, and 3 = unable to do (the worst outcome). Each category is given a score by taking the maximum score of each question (i.e., question in each category with the highest score for that category). The HAQ-DI was calculated by dividing the sum of the category scores by the number of categories with at least 1 question answered.
Time Frame: Core baseline, Week 12
Population: mITT Population Subjects with a missing baseline are not included. Intermediate missing data are imputed using surrounding visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm 1: OKZ 64 mg q4w + MTX | Treatment Arm 2: OKZ 64 mg q2w + MTX
Number analyzed (Participants) | 1057 | 1047
score on a scale
  Core Baseline: number analyzed (Participants) | 1043 | 1022
  Core Baseline | 1.70 (0.581) | 1.74 (0.561)
  Week 12 OLE: number analyzed (Participants) | 1001 | 986
  Week 12 OLE | 1.03 (0.632) | 1.00 (0.628)
  Change from Core Baseline: number analyzed (Participants) | 1001 | 986
  Change from Core Baseline | -0.67 (0.628) | -0.74 (0.648)

14. Secondary Outcome: Change in Health Assessment Questionnaire-Disability Index (HAQ-DI) From Core Baseline at Week 20
Description: as for outcome 13
Time Frame: Core baseline, Week 20
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm 1: OKZ 64 mg q4w + MTX | Treatment Arm 2: OKZ 64 mg q2w + MTX
Number analyzed (Participants) | 1057 | 1047
score on a scale
  Core Baseline: number analyzed (Participants) | 1043 | 1022
  Core Baseline | 1.70 (0.581) | 1.74 (0.561)
  Week 20 OLE: number analyzed (Participants) | 982 | 968
  Week 20 OLE | 1.00 (0.647) | 0.99 (0.621)
  Change from Core Baseline: number analyzed (Participants) | 982 | 968
  Change from Core Baseline | -0.70 (0.631) | -0.74 (0.640)

15. Secondary Outcome: Change in Health Assessment Questionnaire-Disability Index (HAQ-DI) From Core Baseline at Week 28
Description: as for outcome 13
Time Frame: Core baseline, Week 28
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm 1: OKZ 64 mg q4w + MTX | Treatment Arm 2: OKZ 64 mg q2w + MTX
Number analyzed (Participants) | 1057 | 1047
score on a scale
  Core Baseline: number analyzed (Participants) | 1043 | 1022
  Core Baseline | 1.70 (0.581) | 1.74 (0.561)
  Week 28 OLE: number analyzed (Participants) | 955 | 947
  Week 28 OLE | 0.99 (0.632) | 0.99 (0.627)
  Change from Core Baseline: number analyzed (Participants) | 955 | 947
  Change from Core Baseline | -0.71 (0.645) | -0.75 (0.652)

16. Secondary Outcome: Change in Health Assessment Questionnaire-Disability Index (HAQ-DI) From Core Baseline at Week 40
Description: as for outcome 13
Time Frame: Core baseline, Week 40
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm 1: OKZ 64 mg q4w + MTX | Treatment Arm 2: OKZ 64 mg q2w + MTX
Number analyzed (Participants) | 1057 | 1047
score on a scale
  Core Baseline: number analyzed (Participants) | 1043 | 1022
  Core Baseline | 1.70 (0.581) | 1.74 (0.561)
  Week 40 OLE: number analyzed (Participants) | 926 | 917
  Week 40 OLE | 0.97 (0.651) | 0.99 (0.635)
  Change from Core Baseline: number analyzed (Participants) | 926 | 917
  Change from Core Baseline | -0.72 (0.663) | -0.75 (0.672)

17. Secondary Outcome: Change in Health Assessment Questionnaire-Disability Index (HAQ-DI) From Core Baseline at Week 52
Description: as for outcome 13
Time Frame: Core baseline, Week 52
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm 1: OKZ 64 mg q4w + MTX | Treatment Arm 2: OKZ 64 mg q2w + MTX
Number analyzed (Participants) | 1057 | 1047
score on a scale
  Core Baseline: number analyzed (Participants) | 1043 | 1022
  Core Baseline | 1.70 (0.581) | 1.74 (0.561)
  Week 52 OLE: number analyzed (Participants) | 888 | 888
  Week 52 OLE | 0.97 (0.653) | 0.96 (0.623)
  Change from Core Baseline: number analyzed (Participants) | 888 | 888
  Change from Core Baseline | -0.72 (0.670) | -0.77 (0.671)

18. Secondary Outcome: Change in Health Assessment Questionnaire-Disability Index (HAQ-DI) From Core Baseline at Week 64
Description: as for outcome 13
Time Frame: Core baseline, Week 64
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm 1: OKZ 64 mg q4w + MTX | Treatment Arm 2: OKZ 64 mg q2w + MTX
Number analyzed (Participants) | 1057 | 1047
score on a scale
  Core Baseline: number analyzed (Participants) | 1043 | 1022
  Core Baseline | 1.70 (0.581) | 1.74 (0.561)
  Week 64 OLE: number analyzed (Participants) | 876 | 877
  Week 64 OLE | 0.95 (0.641) | 0.97 (0.635)
  Change from Core Baseline: number analyzed (Participants) | 876 | 877
  Change from Core Baseline | -0.74 (0.643) | -0.77 (0.671)

19. Secondary Outcome: Change in Health Assessment Questionnaire-Disability Index (HAQ-DI) From Core Baseline at Week 82
Description: as for outcome 13
Time Frame: Core baseline, Week 82
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm 1: OKZ 64 mg q4w + MTX | Treatment Arm 2: OKZ 64 mg q2w + MTX
Number analyzed (Participants) | 1057 | 1047
score on a scale
  Core Baseline: number analyzed (Participants) | 1043 | 1022
  Core Baseline | 1.70 (0.581) | 1.74 (0.561)
  Week 82 OLE: number analyzed (Participants) | 828 | 855
  Week 82 OLE | 0.97 (0.667) | 0.98 (0.667)
  Change from Core Baseline: number analyzed (Participants) | 828 | 855
  Change from Core Baseline | -0.72 (0.680) | -0.74 (0.695)

20. Secondary Outcome: Proportion of Subjects With Health Assessment Questionnaire - Disability Index (HAQ-DI) Improvement Through Week 82
Description: The number and proportion of subjects with HAQ-DI improvement ≥ 0.22 Against OLE Baseline.
  HAQ-DI Range: 0 (the best outcome) - 3 (the worst outcome), with a decrease from baseline indicating improvement.
  The HAQ-DI assesses the degree of difficulty experienced in 8 domains of daily living activities using 20 questions. The domains are dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities, and each domain (activity) consists of 2 or 3 items. For each question, the level of difficulty is scored from 0 to 3, where 0 = without any difficulty (the best outcome), 1 = with some difficulty, 2 = much difficulty, and 3 = unable to do (the worst outcome). Each category is given a score by taking the maximum score of each question (i.e., question in each category with the highest score for that category). The HAQ-DI was calculated by dividing the sum of the category scores by the number of categories with at least 1 question answered.
Time Frame: up to week 82
Population: Intermediate missing data are imputed using surrounding visits. The OLE Baseline value was defined as the last available measurement prior to the first OLE dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm 1: OKZ 64 mg q4w + MTX | Treatment Arm 2: OKZ 64 mg q2w + MTX
Number analyzed (Participants) | 1057 | 1047
Participants
  Week 12 OLE | 297 | 324
  Week 20 OLE | 319 | 341
  Week 28 OLE | 326 | 320
  Week 40 OLE | 310 | 333
  Week 52 OLE | 322 | 338
  Week 64 OLE | 317 | 326
  Week 82 OLE | 326 | 373

21. Secondary Outcome: Changes From Core Baseline Over Time in Clinical Disease Activity Index (CDAI)
Description: CDAI Range: 0 (the best outcome) - 76 (the worst outcome), with a decrease from baseline indicating improvement.
  The CDAI was calculated in the statistical database for analysis purposes using the SJC (28 joints), TJC (28 joints), the Patient Global Assessment of Disease Activity (VAS) (in cm), and the Physician Global Assessment (VAS) (in cm) according to the following formula: CDAI = SJC + TJC + Patient Global Assessment of Disease Activity (VAS) + Physician Global Assessment (VAS)
Time Frame: up to week 82
Population: Subjects with a missing baseline are not included. Intermediate missing data are imputed using surrounding visits. Baseline is defined as the last available assessment prior to the first dose of the study treatment in the core study.
Measure: Mean (Standard Deviation); unit: index units
Arm/Group | Treatment Arm 1: OKZ 64 mg q4w + MTX | Treatment Arm 2: OKZ 64 mg q2w + MTX
Number analyzed (Participants) | 1057 | 1047
index units
  Core Baseline Actual Values: number analyzed (Participants) | 1014 | 995
  Core Baseline Actual Values | 40.20 (11.252) | 40.06 (11.605)
  Week 12 OLE Actual Values: number analyzed (Participants) | 967 | 953
  Week 12 OLE Actual Values | 10.92 (9.349) | 10.54 (9.106)
  Change from Core Baseline at week 12: number analyzed (Participants) | 967 | 953
  Change from Core Baseline at week 12 | -29.35 (12.093) | -29.54 (12.946)
  Week 20 OLE Actual Values: number analyzed (Participants) | 956 | 943
  Week 20 OLE Actual Values | 10.30 (9.489) | 9.90 (8.755)
  Change from Core Baseline at week 20: number analyzed (Participants) | 956 | 943
  Change from Core Baseline at week 20 | -29.87 (12.553) | -30.23 (12.821)
  Week 28 OLE Actual Values: number analyzed (Participants) | 929 | 922
  Week 28 OLE Actual Values | 9.77 (8.583) | 9.85 (8.696)
  Change from Core Baseline at week 28: number analyzed (Participants) | 929 | 922
  Change from Core Baseline at week 28 | -30.35 (12.111) | -30.36 (12.849)
  Week 40 OLE Actual Values: number analyzed (Participants) | 897 | 891
  Week 40 OLE Actual Values | 9.19 (8.498) | 9.34 (8.235)
  Change from Core Baseline at week 40: number analyzed (Participants) | 897 | 891
  Change from Core Baseline at week 40 | -30.88 (11.992) | -30.80 (13.025)
  Week 52 OLE Actual Values: number analyzed (Participants) | 865 | 865
  Week 52 OLE Actual Values | 8.69 (7.954) | 8.61 (7.776)
  Change from Core Baseline at week 52: number analyzed (Participants) | 865 | 865
  Change from Core Baseline at week 52 | -31.35 (11.855) | -31.60 (12.639)
  Week 64 OLE Actual Values: number analyzed (Participants) | 851 | 853
  Week 64 OLE Actual Values | 8.42 (7.997) | 8.36 (7.798)
  Change from Core Baseline at week 64: number analyzed (Participants) | 851 | 853
  Change from Core Baseline at week 64 | -31.68 (11.896) | -31.85 (12.484)
  Week 82 OLE Actual Values: number analyzed (Participants) | 804 | 829
  Week 82 OLE Actual Values | 9.66 (10.513) | 9.36 (10.236)
  Change from Core Baseline at week 82: number analyzed (Participants) | 804 | 829
  Change from Core Baseline at week 82 | -30.48 (12.878) | -30.58 (14.404)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were reported from OLE Baseline (the same visit as the Week 24 visit in the core studies) until the end of the follow-up period (safety follow-up (SFU-3)). Any AE, including any AE still ongoing at the end of the study, was to be followed until it had resolved, it had a stable sequelae, the Investigator determined that it was no longer clinically significant, or the subject was lost to follow-up.
Description: Safety population consists of all subjects who received at least 1 dose of study treatment during the OLE study CL04041024 . AEs that started before patient enrollment to the OLE study (during core studies CL04041022 (NCT02760368), CL04041023 (NCT02760407) or CL04041025 (NCT02760433) are presented in relevant records for these studies in Clinicaltrials.gov).
Arm/Group | Treatment Arm 1: OKZ 64 mg q4w + MTX | Treatment Arm 2: OKZ 64 mg q2w + MTX
All-Cause Mortality (participants affected / at risk) | 13/1043 | 13/1061
Serious Adverse Events (participants affected / at risk) | 129/1043 | 120/1061
Other Adverse Events (participants affected / at risk) | 356/1043 | 386/1061
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm 1: OKZ 64 mg q4w + MTX (N=1043) | Treatment Arm 2: OKZ 64 mg q2w + MTX (N=1061)
Pneumonia (Infections and infestations) | 7 (7) | 7 (7)
Cellulitis (Infections and infestations) | 7 (7) | 4 (4)
Erysipelas (Infections and infestations) | 5 (5) | 4 (4)
COVID-19 (Infections and infestations) | 1 (1) | 3 (3)
Pyelonephritis acute (Infections and infestations) | 2 (2) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Pyelonephritis (Infections and infestations) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 3 (3)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 1 (1)
Abscess soft tissue (Infections and infestations) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bartholinitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Bullous erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1)
Cat scratch disease (Infections and infestations) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1)
Encephalomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0)
Joint abscess (Infections and infestations) | 1 (1) | 0 (0)
Latent tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Ludwig angina (Infections and infestations) | 1 (1) | 0 (0)
Medical device site abscess (Infections and infestations) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Necrotising soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Renal abscess (Infections and infestations) | 1 (1) | 0 (0)
Salpingo-oophoritis (Infections and infestations) | 1 (1) | 0 (0)
Scrotal abscess (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection pseudomonas (Infections and infestations) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (6)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic intracranial haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary gland calculus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Central nervous system neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 4 (4) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Carotid artery aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Pineal gland cyst (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 7 (7) | 5 (6)
Hepatic enzyme increased (Investigations) | 1 (1) | 1 (1)
Liver function test increased (Investigations) | 1 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1)
Sudden death (General disorders) | 1 (1) | 1 (1)
Lithiasis (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Vascular stent occlusion (General disorders) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Genital haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenic cyst (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Ocular myasthenia (Eye disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm 1: OKZ 64 mg q4w + MTX (N=1043) | Treatment Arm 2: OKZ 64 mg q2w + MTX (N=1061)
Nasopharyngitis (Infections and infestations) | 71 (90) | 87 (108)
Upper respiratory tract infection (Infections and infestations) | 59 (70) | 67 (84)
Bronchitis (Infections and infestations) | 59 (66) | 45 (51)
Alanine aminotransferase increased (Investigations) | 95 (156) | 115 (194)
Aspartate aminotransferase increased (Investigations) | 52 (80) | 63 (94)
Leukopenia (Blood and lymphatic system disorders) | 46 (66) | 60 (95)
Neutropenia (Blood and lymphatic system disorders) | 42 (79) | 57 (92)
Lymphopenia (Blood and lymphatic system disorders) | 41 (62) | 50 (90)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 25 (25) | 42 (44)
Hypertension (Vascular disorders) | 32 (33) | 44 (49)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study related information could be made public available only after Sponsors written permission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/49/NCT03120949/Prot_SAP_000.pdf